CLINICAL TRIAL: NCT02571751
Title: Open-label, Multi-center Trial to Evaluate Safety and Efficacy of Cohesive Silicone Gel-Filled Breast Implants UNIGEL®
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Sewoon Medical Co., Ltd (Industry)
Collaborators: Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol Approval No. 534
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Breast Augmentation

ARMS (1):
- Breast Augmentation (Experimental)
  Interventions: Device: UNIGEL Silicone Gel-Filled Breast Implant

INTERVENTIONS:
Device: UNIGEL Silicone Gel-Filled Breast Implant

SUMMARY:
Open-label, Multi-center, Clinical trial to Evaluate Safety and Efficacy of Cohesive Gel-Filled Breast Implants UNIGEL® Targeting of Women from 22 to 60 Aged with regard to Augmentation Mammaplasty for Purpose of Cosmetic Surgery.

ELIGIBILITY:
Inclusion Criteria:

* Has given written informed consent to entry
* Female, 22 years to 60 years
* Breast augmentation(cosmetic surgery) is for following subjects

  * Who is not content with breast size and shape
  * Who has congenital asymmetrical deformity
* subject who agree to MRI scan during the trial
* subject who agree to visit to hospital according to schedule specified in the protocol during the entire period of the trial

Exclusion Criteria:

* Pregnant or lactating women and women of childbearing age
* Subject who has operation history of breast augmentation or reconstruction
* Subject who has fibrocystic Breast Disease coming up for precancerous lesion not accompanied with subcutaneous mastectomy
* Subject who has breast cancer or prodromal phase and no proper treatment.
* Subject who is diagnosed with Breast Imaging-Reporting and Data System(BI-RADS) category 3 under breast ultrasonography.
* Subject who has uncontrolled active infectious disease or abscess
* Autoimmune disease
* Diabetes mellitus
* Keloidosis
* Subject who cannot take general anesthesia due to abnormal blood or ECG results.
* Subject who is not appropriate for breast augmentation due to damaged tissue or blood vessel or ulcer
* Subject who has metal materials in a body such as ventricular assist system or cerebral aneurysm clips, or has claustrophobia (not suitable for MRI SCAN)
* Physically/mentally disabled subject that may disturb understanding and cooperation for the trial.
* Any other conditions that may interfere with correct assessment of the trial.

Ages: 22 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
a rate of rupture of 4% | 2 years
a rate of capsular contracture of 10% | 2 years

SECONDARY OUTCOMES:
Kaplan-Meier Analysis of rupture or capsular contracture events | 2 years
Change in nipple sensitivity | 2 years
a rate of adverse evnets | 2 years
Change in chest, bust and under bust circumference | 2 years
SF-36(Short Form (36) Health Survey ), Evaluation of quality of life | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea